CLINICAL TRIAL: NCT03674580
Title: Impairment of the Cognitive Flow in the Development of a Depressive Disorder and Suicidal Ideas
Acronym: AQUARIUM
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1515
Record Dates: First submitted 2016-09-13; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Suicide
Keywords: suicidal patients;psychiatry
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suicidal patients: No intervention. Follow-up of the suicidal patients
  Interventions: Behavioral: Follow-up of the suicidal patients

INTERVENTIONS:
Behavioral: Follow-up of the suicidal patients — No intervention. Follow-up of the suicidal patients

SUMMARY:
The study consists in estimating the mental load (cognitive saturation) and the production of driving cognition to suicidal patients.

DETAILED DESCRIPTION:
The study consists in testing two big general hypotheses:

* In the first place, that suicidals presents a mental load (cognitive saturation) and an activity pain behaviour of their space of the thought by extremely painful peripheral cognitive movements (impression that the brain is saturated of thoughts, turbulences, internal movements)
* Secondly, that suicidals produces a surplus of representations of action, such takes out that their vision of the world is saturated of a not integrable kinaesthetic imaging by the subject.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed within the framework of an ambulatory follow-up post-emergencies(post-urgent matters).
* Knowledge of the French language
* patient who have signed of the form of consent,
* patient presenting one anxio-depressive disorder(confusion) with or without suicidal episode.

Exclusion Criteria:

* Not compatible health with the signing of the protocol,
* the not knowledge of the French language,
* patient who have refused the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suicidal patients followed at the Hospital Rene Dubos
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mental load (calm or turbulence of the spirit) - test of the aquarium | 5 days
  To assess the calm or the turbulence of the spirit of the participant, the investigator will make him take the test of the aquarium. The participant will perform an exercise to assess the load and movement of his thoughts. The participant must imagine that the aquarium reflects the content of his mind. The fish are the thoughts and the waves represent the turbulences and movements of all these thoughts. Some subjects, for example, play about with the size of the fish ("it is only a single large fish, but it takes over my entire head"), the shape of the fish ("these fish are pointed because they are bad"), scrawl (the participant scrawled on the aquarium to say that his head was overrun), the projection of feelings ("those fish there are sad") or made digressive but interesting comments ("the wavy lines carry away the fish...").

SECONDARY OUTCOMES:
Moral pain - Analog Visual Scale Battery | 5 days
  In order to evaluate the participant's moral pain, the investigator proposes to answer the questions of a test titled Analog Visual Scale Battery. It is in the form of a horizontal bar with left a peaceful state (mental pain not strong at all...) and conversely, on the right are the opposite feelings corresponding to a moral pain (very strong mental pain). The participant is asked to check on the bar the level that most seems to reflect his feelings or impressions related to his moral pain.
Suicidal thoughts - Analog Visual Scale Battery | 5 days
  In order to evaluate the participant's situation, the investigator proposes to answer the questions of a test titled Analog Visual Scale Battery. It is in the form of a horizontal bar with left a peaceful state (example: calm thoughts, slight suicidal ideation ...) and conversely, on the right are the opposite feelings corresponding to a tormented state (example: many thoughts, suicidal ideation ...). The participant is asked to check on the bar the level that most seems to reflect his feelings or impressions related to his suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: BAUDOIN Thierry, PH, Principal Investigator — Rene Dubos Hospital
Locations (1):
- CH Rene Dubos, Pontoise, Val d'Oise, France

IPD SHARING:
Plan to Share IPD: No